CLINICAL TRIAL: NCT06641804
Title: Effect of Materials of Vaginal Ring Pessary for Pelvic Organ Prolapse on the Effects of Complications and Patient's Satisfaction
Brief Title: Vaginal Prolapse Pessary Material Trial PVC vs Silicon
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Lo Cheuk Yin, Resident, Department of Obstetrics and Gynaecology, Princess Margaret Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pessary material trial
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolpase; ring pessary; silicon ring pessary; PVC ring pessary
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silicon ring pessary (Active Comparator): Change to silicon ring pessary of nearest size
  Interventions: Procedure: Pessary care, change of pessary
- PVC ring pessary (Placebo Comparator): Change of same PVC ring pessary
  Interventions: Procedure: Pessary care, change of pessary

INTERVENTIONS:
Procedure: Pessary care, change of pessary — Insertion of a new pessary by gynaecologist if not contraindicated, silicon or polyvinyl chloride pessary of same size, blinded to patient

SUMMARY:
The goal of this clinical trial is to determine the effect of vaginal ring pessary material on pessary complications and patients' satisfaction.

Participants who are using PVC (polyvinyl chloride) pessary will be randomized to

1. PVC vaginal ring pessary
2. Silicon vaginal ring pessary

Their pessary-related complications, patients' satisfaction, pain during pessary exchange and prolapse related symptoms with reference to PFDI-20 score will be assessed in a period of six months.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a common gynaecological condition which attains prevalence of 15% women. It causes negative impact on physical, emotional and psychosexual aspects, thus significantly impairs patients' activities of daily living and quality of life. Treatment modalities include conservative, pessary and surgical management. Vaginal pessary is inexpensive, non-invasive and an attractive treatment option for women who possess high anaesthetic and surgical risks. Pessary-related complications include vaginal ulcer, vaginitis which would require temporary discontinuation of pessary use in order to prevent serious complications such as incarceration and fistula formation. If complications can be minimised, it is more likely that patients' satisfaction can further improve.

Vaginal pessaries are primarily made of polyvinyl chloride (PVC) or silicone. PVC has been the material of choice for local practice based on its long history in clinical use and cheaper cost. A new PVC pessary is inserted at each consultation if vaginal condition is satisfactory. In view of the increasing number of POP patients who opt for long term pessary use, silicone has emerged as alternative material of choice in recent years. Despite being more expensive, silicone pessaries can be washed and re-inserted for 20 washes/10 years if remained intact and not visibly damaged. As silicone pessary is more pliable, it can facilitate the process of pessary insertion and removal by squeezing of the pessary to pass through narrow introitus. On the other hand, it may be more easily compressed by abdominal pressure and dislodged when straining. The UK clinical guideline for best practice in the use of vaginal pessaries for POP in 2021 suggested there is no clear preference of offering one type of pessary over another, further supported by the latest publication of a multi-centre pessary study in the UK in 2023.

The primary objective is to determine the effect of vaginal ring pessary material on pessary complications and patients' satisfaction. The secondary objectives are to explore the effect of pessary material on procedural pain during pessary exchange as well as prolapse-related symptoms. It is hypothesised that silicone pessaries, compared to PVC pessaries, can reduce the rate of pessary-related complications from 30% to 10% and also result in higher patients' satisfaction.

This is a single-blinded, randomised placebo-controlled trial conducted in the pessary clinic in Princess Margaret Hospital

Participants are assessed for eligibility when they present to pessary clinic for routine pessary care.

Participants are recruited and assigned randomly in 1:1 ratio to receive either

* Treatment arm: replacement of a new silicone pessary
* Control arm: replacement of a new PVC pessary Participants are randomly assigned to one of the two groups in 1:1 ratio. Randomization is carried out by an independent statistician according to computer-generated random numbers in random blocks of two, four and six, allocated by sequentially numbered, sealed opaque envelopes. When participants are prepared for pessary care inside the examination room, the new pessary will be prepared by research assistant outside the examination room according to the allocation result. The attending staff will conduct routine pessary care including pessary removal, vaginal examination and pessary replacement. Participants are not informed of the material of the new pessary. Standard patient information leaflet regarding pessary care with hotlines is provided. A 6-month follow up appointment will be arranged.

Participants will subsequently attend follow up 6 months later. A questionnaire will be given by the research assistant before the consultation to enquire for any pessary-related symptoms, and their satisfaction on the current pessary. During the consultation, the attending staff will remove the study pessary and assess the vaginal condition. The study is concluded by a short questionnaire and routine pessary care follows subsequently.

Data Collection Patient age, parity, menopausal status, stage of prolapse on presentation, previous duration of pessary use, history of pessary complications are obtained from hospital record as demographic data.

Symptoms of pessary-related complications and patients' satisfaction are collected by self-administered questionnaires. Signs of pessary-related complications are assessed and documented by the attending staff.

Statistical Analysis Baseline characteristics and outcomes of PVC pessary group and silicone pessary group are compared using independent t-test, Mann-Whitney U test, Pearson's chi-square test or Fisher's exact test, where appropriate.

Odds ratio for complications with 95% confidence interval was calculated. The within-group changes of patient satisfaction and severity of prolapse with POP-Q were assessed using Wilcoxon signed-rank test.

Sample size calculation Previous pessary study in our unit has shown the rate of pessary-related complications with follow-up interval of 6-month was 30% (only PVC pessary was available) Assuming the complication rate of silicone pessary use with 6-month follow-up interval is 10%, configuring 80% power of detection, 5% of beta error and 20% of dropout rate, 140 participants are needed for recruitment.

ELIGIBILITY:
Inclusion criteria

* At least 18 years old who understand written traditional Chinese
* Diagnosed with stage 1-4 POP according to the standard of Pelvic organ prolapse Quantification (POP-Q)
* Using PVC pessary as long term management for POP
* Willing to participate and provide a written informed consent.

Exclusion criteria

* Do not understand or comprehend written traditional Chinese
* Cannot provide written consent
* Vaginal complication requiring discontinuation of pessary use
* Unable to follow up clinic 6 months later
* Pregnant or lactating
* Recruited in other research studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with vaginal prolapse on pessary care
Enrollment: 140 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pessary related complications | 6 months
  Patient reported symptoms such as vaginal bleeding, vaginal discharge, pessary dislodgement Physician reported complications such as ulcers formation, vaginitis
Patient satisfaction | 6 months
  Visual analogue score 1- 10 [Minimal satisfaction: 1, Maximal satisfaction: 10]

SECONDARY OUTCOMES:
Pain during pessary exchange | 6 months
  Visual analogue scale 1- 10 [Minimal pain: 1, Maximal pain: 10]
Prolapse related symptoms | 6 months
  PFDI 20 summary score (Pelvic Floor Disability Index) [Minimal symptoms: 0 Maximal symptoms: 300]

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk Yin Lo, MBBS, Principal Investigator — Princess Margaret Hospital, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT06641804/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT06641804/ICF_001.pdf